CLINICAL TRIAL: NCT00003688
Title: Pulse Actinomycin-D as Salvage Therapy for Failed Low Risk Gestational Trophoblastic Neoplasia
Brief Title: Dactinomycin in Treating Patients With Persistent or Recurrent Gestational Trophoblastic Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066791; GOG-176
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2003-12

CONDITIONS: Gestational Trophoblastic Tumor
Keywords: recurrent gestational trophoblastic tumor; nonmetastatic gestational trophoblastic tumor; low risk metastatic gestational trophoblastic tumor
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Dactinomycin

INTERVENTIONS:
Biological: dactinomycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dactinomycin in treating patients who have persistent or recurrent gestational trophoblastic neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of dactinomycin in patients with persistent or recurrent low-risk gestational trophoblastic neoplasia.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive dactinomycin IV over 15 minutes on day 1. Treatment repeats every 2 weeks in the absence of unacceptable toxicity. Patients who achieve normal beta-human chorionic gonadotropin (HCG) receive 2 additional courses after attaining normal beta-HCG.

Patients are followed every 2 weeks for 2 months and then monthly for 10 months.

PROJECTED ACCRUAL: A total of 15-35 patients will be accrued for this study within 18-42 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed complete or partial mole on initial evaluation

  * Current diagnosis of persistent or recurrent low-risk gestational trophoblastic neoplasia, defined by 1 of the following criteria:

    * Less than 10% fall in beta-human chorionic gonadotropin (HCG) over 3 consecutive weekly titers
    * More than 20% rise in beta-HCG over the previous value at any time
    * Rise in beta-HCG (greater than 5 mU/mL) after attaining normal level
* Prior treatment limited to methotrexate (MTX) with or without leucovorin calcium (CF)
* WHO score 2-6 at time of relapse
* Must have undergone at least 1 prior curettage for diagnosis and initial management
* No metastatic disease other than lung or vagina on physical examination, chemistry, chest x-ray, or ultrasound
* No more than 8 metastatic lesions
* No histologically confirmed placental site trophoblastic tumor at initial evaluation

PATIENT CHARACTERISTICS:

Age

* 12 to 50

Performance status

* GOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* No significant infection
* No more than 1 year since prior pregnancy
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 1 week since prior chemotherapy and recovered
* No prior chemotherapeutic drugs other than MTX with or without CF

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* Recovered from prior surgery
* No concurrent curettage unless required to control vaginal bleeding

Other

* No prior anticancer treatment that would preclude study therapy

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Covens, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (29):
- United States (28):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Brookview Research, Inc., Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Covens A, Filiaci VL, Burger RA, Osborne R, Chen MD; Gynecologic Oncology Group. Phase II trial of pulse dactinomycin as salvage therapy for failed low-risk gestational trophoblastic neoplasia: a Gynecologic Oncology Group study. Cancer. 2006 Sep 15;107(6):1280-6. doi: 10.1002/cncr.22118. PMID 16900525